CLINICAL TRIAL: NCT03277820
Title: Effect of Probiotics on Microbiome of Adenoid Tissue and Middle Ear Fluid of Children With Otitis Media With Effusion
Brief Title: Effect of Probiotics on Nasopharyngeal Microbiome of Children With Otitis Media With Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, prof. dr. An Boudewyns, MD, PhD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B300201731908
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Otitis Media With Effusion; Probiotics; Adenoid Vegetations
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator does not know which subjects administered probiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Intake of 1 portion (=6 droplets) Probactiol Mini during 4 weeks.
  Interventions: Dietary Supplement: Probactiol Mini
- Control group (No Intervention): No intake of Probactiol Mini

INTERVENTIONS:
Dietary Supplement: Probactiol Mini — 6 droplets of Probactiol Mini contain 1 billion bacteria (Lactobacillus rhamnosus GG and Bifidobacterium lactis BB-12)
  Arms: Probiotic group

SUMMARY:
The aim of this study is to investigate whether the microbiota in the upper respiratory tract (nasopharynx, adenoids and middle ear fluid) of otitis media with effusion (OME) patients is changed after 4 weeks of probiotic product intake. Therefore, bacterial DNA from swabs, fluid and tissue will be isolated via commercially available DNA extraction kits, followed by Illumina MiSeq sequencing in order to identify the bacterial species present in these samples. Furthermore, the concentration of specific pathogens will be monitored via qPCR.

ELIGIBILITY:
Inclusion Criteria:

* children with otitis media with effusion
* children with adenoid hypertrophy

Exclusion Criteria:

* no patients with trisomy 21

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Microbiome differences | 4 years
  After Illumina MiSeq sequencing, bio-informatic tools will be used to cluster bacteria into operational taxonomic units (OTUs). Based on these OTUs, we will compare the composition of the bacteria in the sampled niches and compare this composition between patient with and without intake of probiotics. We will specifically screen for OTUs that are over- or underrepresented in both populations. Furthermore, special attention will go to screen for the typical nasopharyngeal pathogens such as Staphylococcus aureus, Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis... and also to beneficial microbes such as lactic acid bacteria.

SECONDARY OUTCOMES:
Differences in absolute concentration of otitis media pathogens | 4 years
  After DNA extraction of the biological samples, the absolute concentration of the administered probiotics and otitis media pathogens will be monitored via qPCR. This will give information about the capacity of the probiotics to colonise the nasopharynx and to alter the concentration of pathogens.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No